CLINICAL TRIAL: NCT00825669
Title: A Randomized Controlled Trial of Treatment of Portal Vein Tumor Thrombus After Hepatocellular Carcinoma Resection
Brief Title: Treatment of Portal Vein Tumor Thrombus After Hepatocellular Carcinoma Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospotal, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EHBH-RCT-2008-015
Record Dates: First submitted 2009-01-16; First posted 2009-01-21 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; Portal vein tumor thrombus; laser ablation
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- survival rate (TACE) (Active Comparator): to compare the effects of TACE and TACE plus laser ablation for treating patients with PVTT
  Interventions: Drug: TACE
- survival rate (TACE plus laser ablation) (Active Comparator): to compare the effects of TACE and TACE plus laser ablation for treating patients with PVTT
  Interventions: Drug: TACE; Procedure: Laser ablation

INTERVENTIONS:
Drug: TACE — TACE: The chemotherapeutic drugs and 2 to 10 ml lipiodol are given via hepatica propria artery. The chemotherapeutic drugs include 5-Fu 1500 mg, epirubicin 30 mg, cisplatin 30 mg.
  Other Names: TAE
Procedure: Laser ablation — Laser ablation is given to the PVTT.
  Other Names: Microinvasive
  Arms: survival rate (TACE plus laser ablation)

SUMMARY:
Hepatectomy is still the treatment of choice for hepatocellular carcinoma. Part of the patients may present portal vein tumor thrombus (PVTT) after resection. PVTT might lead to upper gastrointestinal bleeding and worsening of hypersplenism which will endanger the life of the patients. PVTT also plays the centre role of recurrence and metastasis of HCC. There is no standard treatment for PVTT yet. We aim to compare the effects of TACE and TACE plus laser ablation for treating patients with PVTT.

DETAILED DESCRIPTION:
Hepatectomy is still the treatment of choice for hepatocellular carcinoma, but the prognosis is not agreeable. Part of the patients may present portal vein tumor thrombus (PVTT) after resection. PVTT might further increase the pressure of portal vein and lead to upper gastrointestinal bleeding and worsening of hypersplenism which will endanger the life of the patients. PVTT also plays the centre role of recurrence and metastasis of HCC. There is no standard treatment available now for PVTT yet. TACE is mostly often used to treat the PVTT. We aim to compare the effects of TACE and TACE plus laser ablation for treating patients with PVTT.

ELIGIBILITY:
Inclusion Criteria:

1. PVTT after liver resection was diagnosed with at least two types of imaging findings, such as CT, MRI or color doplor findings.
2. The functions of the kidney, heart and lung and the routine test of the blood are in good condition.
3. The liver function is of grade A or B in Child-Pugh classification.
4. The patient is eligible of the trial and will show consent to the test.

Exclusion Criteria:

1. any of the parameters. WBC less than 2000/ml, Hb less than 90g/L or PLT less than 50000/ml.
2. disfunction of the heart, lung, kidney, or brain.
3. any other disease might affect the trial .
4. the patients would not sign the consent to the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
overall survival | 2010

SECONDARY OUTCOMES:
the changes of the PVTT | 2010

CONTACTS AND LOCATIONS:
Overall Officials: shen feng, M.D, Study Chair — Eastern Hepatobiliary Surgery Hospital Affiliated to Second Military Medical University
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality, China